CLINICAL TRIAL: NCT06699264
Title: Effekte Von Blood Flow Restriction Therapie Auf Das Schmerzempfinden Bei Patienten Mit Rekonstruktion Des Vorderen Kreuzbandes (Effects of Blood Flow Restriction Therapy on Pain Sensation in Patients With Anterior Cruciate Ligament Reconstruction)
Brief Title: Effects of Low-intensity Strength Training With Concomitant Blood Flow Restriction on Pain Perception in Patients With Anterior Cruciate Ligament Surgery
Acronym: BFR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Praxisklinik Rennbahn AG (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-00151; Forschungsförderung Nr. 106 (Other Grant/Funding Number: Gesellschaft für Arthroskopie und Gelenkchirurgie)
Record Dates: First submitted 2024-11-13; First posted 2024-11-21 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Anterior Cruciate Ligament Injury
Keywords: ACL injury; BFR; Blood flow restriction; Physiotherapy
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): Group 1 (experimental group) will be trained with the intervention method (low-load strength training) using the Tourniquet Touch (VBM Medizintechnik GmbH Einsteinstrasse 1, 72172 Sulz a.N., Germany)
  Interventions: Other: Blood Flow Restriction Training
- Control Group (Active Comparator): Group 2 (controll group) receives the same strength training only without simultaneous restriction blood flow.
  Interventions: Other: Training without BFR

INTERVENTIONS:
Other: Blood Flow Restriction Training — Pressure cuff is applied to the leg during training for low-load strength training with simultaneous restiction of blood flow
  Arms: Experimental Group
Other: Training without BFR — Strength training according to experimentral group without simultaneous restriction blood flow
  Arms: Control Group

SUMMARY:
After surgical treatment of a tear of the anterior cruciate ligament, physiotherapeutic exercises are done as standard therapy. This is to achieve a rapid improvement in pain and knee function. In this study, the Investigators examine how low-intensity strength training with simultaneous restriction of blood flow works and whether it is effective and well tolerated. For this purpose, a pressure cuff is applied to the leg during training. Participation in this study will last four weeks for each participant. The Investigators will invite participants for 11 study visits. One appointment will last about 30 minutes. If a participant decides to take part in the study, they will be randomly assigned to one of two groups. The participants will belong to either an experimental group or the control group. In the experimental group, the participants will be treated with the intervention method. The intervention method involves 4 weeks of low-intensity strength training with an additional pressure cuff on the leg, which should lead to improved adaptations to the muscle as well as a reduction in pain. In the control group, the participants will receive the same strength training only without the additional pressure cuff. The benefit is that in addition to the participants actual rehabilitation program, each participant will receive free training to build their muscles. This could contribute to an accelerated rehabilitation process and a faster build-up of strength as well as an improvement in pain. It is additionally possible that the participants will help future patients with their participation. The intervention method for strength training with simultaneous restriction of blood flow (Blood Flow Restriction Training) has been studied for some time. There is good evidence of improved muscle, tendon and pain adaptations in both healthy individuals and patients with ACL injury. Whether this training method also has an effect on pain perception will be investigated in this study.

Participants may experience side effects if they are treated with the intervention method (low-intensity strength training with simultaneous restriction of blood flow). The Investigators may not yet know all the risks and side effects of the intervention method. So far, the following risks and side effects are known:

* Temporay numbness
* Muscle soreness
* Pressure sensation

ELIGIBILITY:
Inclusion Criteria:

* It must be your first anterior cruciate ligament surgery
* You must be between 18 and 60 years old
* You must be able to successfully complete certain exercises
* The injury must have occurred no longer than 6 months ago

Exclusion Criteria:

* Injury in other ligaments in the knee and cartilage
* thrombosis
* infection
* high blood pressure (which is not treated with medication)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-12-21 (Actual); Study Completion 2024-12-21 (Actual)

PRIMARY OUTCOMES:
Rate of Pressure and Pain Treshold (Wagner FPX) | Pre and post training as well as in week 1 of training
  The Wagner FPX (Wagner Instruments, Greenwich, CT 06836-1217 USA) is used to quantify and document sensitivity and pain thresholds through defined application of pressure. Pain sensitivity is measured in kgf/s at four pre-defined positions:
  Position 1: dominant quadriceps muscles - centered on the muscle belly, 20 cm proximal to the proximal end of the patella Position 2: non-dominant quadriceps muscles - centered on the muscle belly, 20cm proximal to the proximal end of the patella Position 3: dominant m. biceps brachii - centered on the muscle belly, 10 cm proximal to the cubital fossa (= elbow bend) Position 4: non-dominant trapezius muscle (based on handedness) - centered on the muscle belly, 10 cm from the proximal end of the acromion in a direct line to the neck

SECONDARY OUTCOMES:
Legpress 10-repition maximum voluntary contraction test (HUMAC NORM Isokinetic Dynamometer By CSMi) | pre and post training as well as in weeks 3 to 9
  Lower extremity MVC is measured using the HUMAC NORM Isokinetic Dynamometer By CSMi (CSMi, Stoughton, MA 02072, United States) in Nm during a 90° knee-bend legpress. Participants perform 10 repitions with maximum force.
Rate of muscle thickness of the m. rectus femoris in mm | Pre- and post training period
  The muscle thickness of the m. rectus femoris is measured using an ultrasound device (Esaote MyLab Touch, Esaote SPA Genova GE, Italy)

CONTACTS AND LOCATIONS:
Locations (1):
- Praxisklinik Rennbahn AG, Muttenz, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Sensitive Patient Data